CLINICAL TRIAL: NCT01929863
Title: A Randomized, Double-blind (Sponsor Unblinded), Placebo Controlled, Repeat Dose Study Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2330672 in Type 2 Diabetes Patients Taking Metformin
Brief Title: Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2330672 in Type 2 Diabetes Patients Taking Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Elite Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200185
Record Dates: First submitted 2013-08-22; First posted 2013-08-28 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metformin; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Subjects will receive metformin 850 mg BID for 7 days, GSK2330672 45 mg BID on Days 1 and 2 and GSK2330672 90 mg BID on Days 3 to 7 in treatment period 1. Subjects will receive metformin 850 mg BID for 7 days, placebo (matching 45 mg GSK2330672) BID on Days 1 and 2 and placebo (matching 90 mg GSK2330672) BID on Days 3 to 7 in treatment period 2. Treatment periods will be separated by a washout period of 13 to 15 days in which subjects will continue metformin 850 mg BID only
  Interventions: Drug: GSK2330672; Drug: Placebo; Drug: Metformin
- Arm B (Experimental): Subjects will receive metformin 850 mg BID for 7 days, placebo (matching 45 mg GSK2330672) BID on Days 1 and 2 and placebo (matching 90 mg GSK2330672) BID on Days 3 to 7 in treatment period 1. Subjects will receive metformin 850 mg BID for 7 days, GSK2330672 45 mg BID on Days 1 and 2 and GSK2330672 90 mg BID on Days 3 to 7 in treatment period 2. Treatment periods will be separated by a washout period of 13 to 15 days in which subjects will continue metformin 850 mg BID only
  Interventions: Drug: GSK2330672; Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: GSK2330672 — GSK2330672 will be supplied as oral solution, and will be administered BID [45 mg (2 days repeat dose) and 90 mg (5 days repeat dose) in each period]
Drug: Placebo — GSK2330672 matching placebo will be supplied as oral solution, and will be administered BID (7 days of dosing in each period)
Drug: Metformin — Metformin 850 mg will be administered BID from Run-in period till Day 7 of period 2

SUMMARY:
Metformin may have complex interactions in the gut and is generally first line therapy for type 2 diabetes mellitus (T2DM). It is important to understand whether there are significant pharmacokinetic or pharmacodynamic interactions when GSK2330672 is co-administered with metformin in subjects with T2DM. The purpose of this study is to investigate the safety and tolerability of GSK2330672 administered for 7 days to subjects with T2DM taking metformin. This will be a two-period crossover study; subjects will receive either GSK2330672 or placebo for 7 days in each period separated by a washout period of 13 to 15 days. All subjects will receive metformin throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 30 and 64 years of age inclusive, at the time of signing the informed consent.
* Subjects with documented T2DM diagnosis (diagnosed not less than 3 months prior to screening); AND one of the following: taking stable metformin 850 milligrams (mg) twice daily (BID) (or the equivalent of 1700 mg/day) for at least 4 weeks prior to screening and a glycosolated haemoglobin A1c (HbA1c) of >=7.0% to <=11% at screening; OR taking stable metformin of >=1000 mg/day to <1700 mg/day for at least 4 weeks prior to screening and a HbA1c of >=7.5% to <=11% at Screening; OR taking stable metformin of >1700 to <=2000 mg/day for at least 4 weeks prior to screening and a HbA1c of >=7.0% to <=10% at screening; not taking other anti-diabetic medications.
* All T2DM subjects must meet label recommendations for metformin, including: Adequate renal function, as evidenced by the Modification of Diet in Renal Disease estimate of glomerular filtration rate >=60 milliliters (mL)/minute (min); No conditions which make hypoxia, dehydration, or sepsis likely; No clinical or laboratory evidence of hepatic disease (including history of cholecystitis or symptomatic gallstones) and cardiac disease (including a history of myocardial infarction or heart failure). Subjects with a history of cholelithiasis and uncomplicated cholecystectomy more than 3 months before screening may be eligible if approved by the GlaxoSmithKline (GSK) Medical Monitor; No excessive alcohol intake.
* C-peptide of >0.8 nanogram (ng)/mL at screening visit.
* Urine albumin-to-creatinine ratio <30 mg/gram (g).
* Fasting plasma glucose <280 mg/decilitre (dL)
* Body mass index (BMI) of 24 to 40 kilograms (kg)/square meter (m^2), inclusive
* In good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination that would introduce additional risk factors or interfere with study procedures or objectives, based on a medical evaluation including medical history, physical examination, vital signs and laboratory tests.
* Female subjects of non-childbearing potential. Non-childbearing potential is defined as: Pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]. Postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli international units (MIU)/mL and estradiol < 40 picograms (pg)/mL (<147 picomole [pmol]/liter [L]) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the acceptable contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Male subjects with female partners of child-bearing potential must agree to use one of the acceptable contraception methods. This criterion must be followed from the time of the first dose of study medication until follow up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* CRITERIA BASED UPON MEDICAL HISTORIES:
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* History of chronic or acute pancreatitis. Approval from the GSK Medical Monitor must be obtained for subjects with a past history of pancreatitis more than 12 months from the start of the treatment period (subjects with a history of pancreatitis within 12 months prior to the start of the treatment period are excluded).
* History of gastrointestinal (GI) disease (e.g., irritable bowel disease, chronic or current diarrhea, inflamed bowel, steatorrhoea/fat malabsorption, celiac disease, symptomatic lactose intolerance). Subjects with gastroparesis requiring treatment are excluded.
* History of significant cardiovascular disease including acute myocardial infarction, stroke, hospitalization for acute coronary syndrome, heart failure within the previous 12 months.
* Uncontrolled hypertension, as evidenced by systolic pressure >160 or diastolic pressure >90. Subjects taking anti-hypertensive medications are permitted.
* Significant ECG abnormalities, defined as follows: Heart rate (resting) <50 and >100 beats per minute (bpm); PR Interval <120 and >220 milliseconds (msec); QRS duration <70 and >120 msec
* History of untreated pernicious anemia or who have laboratory parameters suggestive of subclinical megaloblastic anemia (e.g., increased mean corpuscular volume with low red blood cells count and/or haemoglobin level).
* Current or relevant previous significant medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that, in the opinion of the investigator, presents undue risk from the study medication or procedures.
* Thyroid Disease: Uncorrected Thyroid Dysfunction: Fasting plasma thyroid stimulating hormone (TSH) outside of the normal range, as determined at the screening visit; Subjects on stable thyroid replacement therapy and with TSH in the normal range are eligible if approved by the GSK Medical Monitor; Unevaluated thyroid nodule or goiter at Screening.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* CRITERIA BASED UPON DIAGNOSTIC ASSESSMENTS:
* Alanine transaminase, alkaline phosphatase and bilirubin > 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on averaged QTcF values of triplicate ECGs obtained at least 1 minute apart within approximately 15 minutes: QTcF >=450 msec; or QTcF >=480 msec in subjects with Bundle Branch Block (subjects with left bundle branch block are excluded)
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for human immunodeficiency virus antibody
* A positive pre-study drug/alcohol urine screen
* A subject with a positive urine cotinine test result will be excluded from the study unless in the judgment of the Investigator the subject will be able to abstain from using tobacco for the duration of the in-house periods of the study.
* OTHER CRITERIA
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* A subject with a fasting plasma glucose at Day -1 that is more than 100 mg/dL lower than at screening must not be randomized, unless on a repeat test the value less than 100 mg/dL of the screening value.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08-01; Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200185 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 16 participants with Type 2 diabetes mellitus (T2DM), aged 30 to 64 years, at a single center of United States from 22 August 2013 to 21 November 2013.
Pre-assignment Details: A total of 15 participants were randomized in the study and entered a run-in period where participants were administered oral dose of metformin 850 milligram (mg) tablet twice daily (BID) for 14 days, after which they entered the 2 double blind treatment periods in a crossover manner.
Groups:
- Metformin and GSK2330672, Then Placebo and Metformin: Participants received oral dose of treatment A-metformin 850 mg BID tablet for 7 days plus GSK2330672 45 mg tablet BID on Day 1 and 2 and GSK2330672 90 mg tablet BID on Day 3 to 7 according to a plan of randomization. After a washout period of 13 to 15 days, participants received oral dose of treatment B-metformin 850 mg tablet BID plus matching placebo to GSK2330672 tablet BID for 7 days. During the washout period, participants received metformin 850 mg tablet BID. After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
- Placebo and Metformin, Then Metformin and GSK2330672: Participants received oral dose of treatment B-metformin 850 mg tablet BID plus matching placebo to GSK2330672 tablet BID for 7 days according to a plan of randomization. After a washout period of 13 to 15 days, participants received oral dose of treatment A-metformin 850 mg BID tablet for 7 days plus GSK2330672 45 mg tablet BID on Day 1 and 2 and GSK2330672 90 mg tablet BID on Day 3 to 7. During the washout period, participants received metformin 850 mg tablet BID. After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
Period: Period 1:Intervention Period 1 (7 Days)
Arm/Group | Metformin and GSK2330672, Then Placebo and Metformin | Placebo and Metformin, Then Metformin and GSK2330672
Started | 7 | 8
Completed | 6 | 7
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2:Washout Period (13-15 Days)
Arm/Group | Metformin and GSK2330672, Then Placebo and Metformin | Placebo and Metformin, Then Metformin and GSK2330672
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Period 3:Intervention Period 2 (7 Days)
Arm/Group | Metformin and GSK2330672, Then Placebo and Metformin | Placebo and Metformin, Then Metformin and GSK2330672
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 4:Follow-up-Metformin (7-10 Days)
Arm/Group | Metformin and GSK2330672, Then Placebo and Metformin | Placebo and Metformin, Then Metformin and GSK2330672
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: In each treatment period, participants received oral dose of treatment A-metformin 850 mg BID tablet for 7 days plus GSK2330672 45 mg tablet BID on Day 1 and 2 and GSK2330672 90 mg tablet BID on Day 3 to 7 or oral dose of treatment B-metformin 850 mg tablet BID plus matchig placebo to GSK2330672 tablet BID for 7 days according to a plan of randomization. The two treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID. After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE), Serious Adverse Event (SAE) or Death
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase (ALT) >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalized ratio >1.5.
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population was defined as all participants enrolled into the study who have received at least one dose of study drug (including metformin, GSK2330672, and matching placebo. One participant withdrew consent after taking period 1 study treatment of placebo + GSK2330672.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A-GSK2330672 + Metformin: Participants received oral dose of metformin 850 mg BID tablet for 7 days plus GSK2330672 45 mg tablet BID on Day 1 and 2 and GSK2330672 90 mg tablet BID on Day 3 to 7 in a sequence of treatment A/B or B/A according to a plan of randomization. Treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID. After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
- Treatment B-Placebo + Metformin: Participants received oral dose of metformin 850 mg tablet BID for 7 days plus matching placebo to GSK2330672 tablet BID for 7 days in a sequence of treatment A/B or B/A according to a plan of randomization. Treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID. After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 14 | 14
Participants
  Any AE | 12 | 9
  Any SAE | 1 | 0
  Any Death | 0 | 0

2. Primary Outcome: Number of Participants With the Indicated Clinical Chemistry Values of Potential Clinical Importance (PCI) at Any Time Post Baseline
Description: The assessments were done at Day -1, Day 3, Day 8 and Follow-up under fasting condition. The following laboratory parameters of clinical chemistry were analyzed: blood urea nitrogen (BUN), creatinine, fasting triglycerides (TGs), total cholesterol, low-density lipoprotein cholesterol (LDLc), high-density lipoprotein cholesterol (HDLc), sodium, potassium, chloride, total bicarbonate, calcium, aspartate aminotransferase (AST), ALT, gamma glutamyltransferase (GGT), alkaline phosphatase, total and direct bilirubin, uric acid, albumin and total protein. Baseline was the assessment done on Day -1 (pre dose). Only those parameters for which at least one value of PCI was reported are summarized. Data is reported for participants with high glucose PCI, where the PCI value for T2DM participants was ( low < 3.8857 millimole per liter (mmol/L); high > 15 mmol/L; normal range was 3.61 - 5.5 mmol/L).
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A-GSK2330672 + Metformin: Participants received oral dose of metformin 850 mg BID tablet for 7 days plus GSK2330672 45 mg tablet BID on Day 1 and 2 and GSK2330672 90 mg tablet BID on Day 3 to 7 in a sequence of treatment A/B or B/A according to a plan of randomization. Treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID.
- Treatment B-Placebo + Metformin: Participants received oral dose of metformin 850 mg tablet BID for 7 days plus matching placebo to GSK2330672 tablet BID for 7 days in a sequence of treatment A/B or B/A according to a plan of randomization. Treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID.
- Follow-up-Metformin: After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Participants | 0 | 0 | 2

3. Primary Outcome: Number of Participants With the Indicated Haematology Values of PCI at Any Time Post Baseline
Description: The assessments were done at Day -1, Day 3, Day 8 and Follow-up under fasting condition. The following laboratory parameters of clinical haematology were analyzed: platelet count, red blood cells (RBC) count, absolute white blood cells (WBC) count, reticulocyte count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline was the assessment done on Day -1 (pre dose). Only those parameters for which at least one value of PCI was reported are summarized. Data is reported for participants with high WBC counts PCI, where the PCI value for T2DM participants was (relative low : 0.5 multiplier of lower limit of normal [LLN]; relative high : 1.82 multiplier of upper limit of normal [LLN]; where normal range was 3.8 - 10.8 giga cells per liter (GI/L).
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Participants | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Values of Urine Microscopic Analysis of Bacteria, Hyaline Casts (Semi-quantitive), RBC, Squamous Epithelial Cells and WBC at Any Time Post Baseline
Description: The assessments were done at Day -1, Day 3, Day 8 and Follow-up under fasting condition for microscopic analysis of bacteria, hyaline casts (semi-quantitive), RBC, squamous epithelial cells and WBC. Baseline was the assessment done on Day -1 (pre dose). The participants were categorized as 0-5, 6-10, 10-20, moderate, few and many. Only those parameters for which at least one value of these categories reported are summarized.
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Participants
  Urine Microscopy, Bacteria, Day 3, Few: number analyzed (Participants) | 14 | 14 | 0
  Urine Microscopy, Bacteria, Day 3, Few | 0 | 1 |
  Urine Microscopy, Bacteria, Day 3, Many: number analyzed (Participants) | 14 | 14 | 0
  Urine Microscopy, Bacteria, Day 3, Many | 0 | 1 |
  Urine Microscopy, Bacteria, Day 8, Few: number analyzed (Participants) | 14 | 14 | 0
  Urine Microscopy, Bacteria, Day 8, Few | 1 | 1 |
  Urine Microscopy, Bacteria, Follow-up, Many: number analyzed (Participants) | 0 | 0 | 15
  Urine Microscopy, Bacteria, Follow-up, Many |  |  | 1
  Urine Microscopy, SEC's, Day 3, 0-5: number analyzed (Participants) | 14 | 14 | 0
  Urine Microscopy, SEC's, Day 3, 0-5 | 0 | 1 |
  Urine Microscopy, SEC's, Day 8, 0-5: number analyzed (Participants) | 14 | 14 | 0
  Urine Microscopy, SEC's, Day 8, 0-5 | 0 | 1 |
  Urine Microscopy, SEC's, Follow-up, 0-5: number analyzed (Participants) | 0 | 0 | 15
  Urine Microscopy, SEC's, Follow-up, 0-5 |  |  | 1
  Urine Microscopy, SEC's, Follow-up, 6-10: number analyzed (Participants) | 0 | 0 | 15
  Urine Microscopy, SEC's, Follow-up, 6-10 |  |  | 1
  Urine Microscopy, WBC's, Day 3, 10-20: number analyzed (Participants) | 14 | 14 | 0
  Urine Microscopy, WBC's, Day 3, 10-20 | 0 | 1 |
  Urine Microscopy, WBC's, Follow-up, 0-5: number analyzed (Participants) | 0 | 0 | 15
  Urine Microscopy, WBC's, Follow-up, 0-5 |  |  | 1
  Urine Microscopy, WBC's, Follow-up, 6-10: number analyzed (Participants) | 0 | 0 | 15
  Urine Microscopy, WBC's, Follow-up, 6-10 |  |  | 1

5. Primary Outcome: Number of Participants With Abnormal Values of Urine Dipstic Analysis of Occult Blood, Glucose, Ketones and Proteins at Any Visit Post Baseline
Description: The assessments were done at Day -1, Day 3, Day 8 and Follow-up under fasting condition for urine dipstic analysis of occult blood, glucose, ketones and proteins. Baseline was the assessment done on Day -1 (pre dose). The participants were categorized with results of 1+, 2+, 3+ and trace. Only those parameters for which at least one value of these categories reported are summarized.
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Participants
  Urine Glucose, Day 3, 1+: number analyzed (Participants) | 14 | 14 | 0
  Urine Glucose, Day 3, 1+ | 1 | 3 |
  Urine Glucose, Day 3, 2+: number analyzed (Participants) | 14 | 14 | 0
  Urine Glucose, Day 3, 2+ | 1 | 0 |
  Urine Glucose, Day 3, Trace: number analyzed (Participants) | 14 | 14 | 0
  Urine Glucose, Day 3, Trace | 1 | 1 |
  Urine Glucose, Day 8, 2+: number analyzed (Participants) | 14 | 14 | 0
  Urine Glucose, Day 8, 2+ | 1 | 3 |
  Urine Glucose, Day 8, Trace: number analyzed (Participants) | 14 | 14 | 0
  Urine Glucose, Day 8, Trace | 2 | 5 |
  Urine Glucose, Follow-up, 3+: number analyzed (Participants) | 0 | 0 | 15
  Urine Glucose, Follow-up, 3+ |  |  | 3
  Urine Glucose, Follow-up, Trace: number analyzed (Participants) | 0 | 0 | 15
  Urine Glucose, Follow-up, Trace |  |  | 3
  Urine Ketones, Day 3, Trace: number analyzed (Participants) | 14 | 14 | 0
  Urine Ketones, Day 3, Trace | 1 | 0 |
  Urine Ketones, Follow-up, Trace: number analyzed (Participants) | 0 | 0 | 15
  Urine Ketones, Follow-up, Trace |  |  | 2
  Urine Protein, Follow-up, Trace: number analyzed (Participants) | 0 | 0 | 15
  Urine Protein, Follow-up, Trace |  |  | 1

6. Primary Outcome: Mean Specific Gravity of Urine at Any Visit Post Baseline
Description: Urine specific gravity is a laboratory test that shows the concentration of all chemical particles in the urine. The assessments were done at Day -1, Day 3, Day 8 and Follow-up under fasting condition. Baseline was the assessment done on Day -1 (pre dose).
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Ratio
  Day 3: number analyzed (Participants) | 13 | 14 | 0
  Day 3 | 1.0121 (0.00352) | 1.0110 (0.00335) |
  Day 8: number analyzed (Participants) | 12 | 14 | 0
  Day 8 | 1.0125 (0.00654) | 1.0109 (0.00386) |
  Follow-up: number analyzed (Participants) | 0 | 0 | 15
  Follow-up |  |  | 1.0203 (0.00832)

7. Primary Outcome: Number of Participants With Abnormal Results for Fecal Occult Blood Test
Description: The assessment of fecal occult blood was done on Day 8. Stool sample was obtained any time after dosing on Day 7.
Time Frame: Day 8 of both treatment periods
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B-Placebo + Metformin: Participants received oral dose of metformin 850 mg tablet BID for 7 days plus matchig placebo to GSK2330672 tablet BID for 7 days in a sequence of treatment A/B or B/A according to a plan of randomization. Treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID. After completion of the double blind treatment period 2 (after the last dose of period 2), participants received oral dose of metformin 850 mg tablet BID for 7-10 days of Follow-up.
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

8. Primary Outcome: Number of Participants With Vital Sign Values of PCI at Any Time Post Baseline
Description: Vital signs assessment included heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP). Assessments were completed at pre morning dose on Day 1 (Baseline), Day 3, Day 8 (before discharge) and Follow-up. Criteria for vital sign values meeting PCI for Type 2 diabetes mellitus (T2DM) included: SBP <85 and >160 millimeters of mercury (mmHg), DBP <45 and >100 mmHg and HR <40 and >110 beats per minute (bpm). Only those parameters for which at least one value of PCI was reported are summarized.
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B-Placebo + Metformin: Participants received oral dose of metformin 850 mg tablet BID for 7 days plus matchig placebo to GSK2330672 tablet BID for 7 days in a sequence of treatment A/B or B/A according to a plan of randomization. Treatment periods were separated by a washout period of 13 to 15 days in which participants continued metformin 850 mg tablet BID.
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Participants
  SBP | 0 | 1 | 0
  HR | 1 | 0 | 0

9. Primary Outcome: Number of Participants With Abnormal (Clinically Significant or Not Clinically Significant) Findings in 12-lead Electrocardiogram (ECG) at Any Time Post Baseline
Description: 12-lead ECG assessments were obtained pre-dose at Day 1, Day 3, Day 8 (before discharge) and Follow-up. The assessments were done using an ECG machine that automatically calculated the heart rate and measures PQ, QRS, QT, and QTc(B) intervals. Abnormal ECG findings (clinically significant or not clinically significant) were categorized. The abnormal PCI range for T2DM participants include QTc interval of >450 to <=480 milliseconds (msec) and increase from Baseline QTc interval of > 30 to <=60 msec, PR interval <110 and >220 msec and QRS interval <75 and >110 msec. ECG abnormalities were categorized as clinically significant or not clinically significant based on PCI criteria and judgment of the investigator. Baseline was defined as the mean of three replicate assessments at pre-dose on Day 1.
Time Frame: Up to Follow-up (up to 53 days)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin | Follow-up-Metformin
Number analyzed (Participants) | 14 | 14 | 15
Participants
  Not-clinically Significant, Day 3: number analyzed (Participants) | 13 | 14 | 0
  Not-clinically Significant, Day 3 | 3 | 2 |
  Clinically Significant, Day 3: number analyzed (Participants) | 13 | 14 | 0
  Clinically Significant, Day 3 | 0 | 0 |
  Not-clinically Significant, Day 8: number analyzed (Participants) | 12 | 14 | 0
  Not-clinically Significant, Day 8 | 2 | 4 |
  Clinically Significant, Day 8: number analyzed (Participants) | 12 | 14 | 0
  Clinically Significant, Day 8 | 0 | 0 |
  Not-clinically Significant, Follow-up: number analyzed (Participants) | 0 | 0 | 15
  Not-clinically Significant, Follow-up |  |  | 3
  Clinically Significant, Follow-up: number analyzed (Participants) | 0 | 0 | 15
  Clinically Significant, Follow-up |  |  | 0

10. Primary Outcome: Number of Events of Stool or Bowel Movements of Participants Using Bristol Stool Form Rating (BSFR) Scale Across Day 1 to 7
Description: The BSFR Scale assessed stool quality using a 7-point scale, where 1=separate hard lumps like nuts (difficult to pass) and 7=watery, no solid pieces (entirely liquid). Bristol Stool Form Scale Rating: 1=separate hard lumps, like nuts, 2=sausage shaped but lumpy, 3=like a sausage or snake but with cracks on its surface, 4=like a sausage or snake, smooth and soft, 5=soft blobs with clear cut edges, 6=fluffy pieces with ragged edges, a mushy stool, 7=watery, no solid pieces. Data is reported for number of events in participants with each category of BSFR scale across Day 1 to 7 post morning dose.
Time Frame: Day 1 to 7 of each treatment period
Population: Safety Population.
Measure: Number; unit: Number of events
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 14 | 14
Number of events
  Participants with Rating 1 | 0 | 6
  Participants with Rating 2 | 4 | 4
  Participants with Rating 3 | 4 | 8
  Participants with Rating 4 | 11 | 20
  Participants with Rating 5 | 18 | 15
  Participants with Rating 6 | 60 | 17
  Participants with Rating 7 | 111 | 16

11. Primary Outcome: Number of Participants in Each Category of BSFR Across Day 1 to 7
Description: The BSFR Scale assessed stool quality using a 7-point scale, where 1=separate hard lumps like nuts (difficult to pass) and 7 = watery, no solid pieces (entirely liquid). Bristol Stool Form Scale Rating: 1=separate hard lumps, like nuts, 2=sausage shaped but lumpy, 3=like a sausage or snake but with cracks on its surface, 4=like a sausage or snake, smooth and soft, 5=soft blobs with clear cut edges, 6=fluffy pieces with ragged edges, a mushy stool, 7=watery, no solid pieces. Data is reported for number of events in participants with each category of BSFR scale across Day 1 to 7 post morning dose.
Time Frame: Day 1 to 7 of each treatment period
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 14 | 14
Participants
  Rating 1 | 0 | 4
  Rating 2 | 3 | 3
  Rating 3 | 4 | 6
  Rating 4 | 5 | 10
  Rating 5 | 8 | 6
  Rating 6 | 12 | 8
  Rating 7 | 14 | 6

12. Primary Outcome: Mean Change From Baseline in Overall Gastrointestinal Symptom Rating Scale (GSRS) Scores
Description: The impact of gastrointestinal (GI) symptoms on health-related quality of life was assessed using the GSRS. The GSRS is a 15-item related to abdominal pain, reflux, indigestion, diarrhea and constipation syndromes, self-administered questionnaire that assesses the impact of gastrointestinal symptoms during the past week on a scale from 1 (no discomfort at all) to 7 (very severe discomfort). Overall GSRS is the mean of questions 1-15 and range from 1 to 7, with lower scores indicating a better quality of life with respect to gastrointestinal symptoms. Baseline was defined as the assessment done on Day -1. Change from baseline was calculated by subtracting the baseline (Day -1) values from the post-baseline value (Day 8).
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 12 | 14
Score on scale | 0.59 (0.891) | 0.08 (0.468)

13. Secondary Outcome: Maximum and Weighted Mean Change From Baseline in Plasma Glucose Concentrations Over a 24 Hour (h) Period on Day 7
Description: Baseline was defined as the time matched assessment done on Day -1. Change from baseline was calculated by subtracting the baseline (Day -1) time matched values from the post-baseline value (Day 8). Data is reported for fasting glucose level and for weighted mean and maximum values for fasting, 0-4 h, 4-10 h, 10-14 h and 0-24 h. Area under the curve (AUC) with respect to these time interval was calculated using the linear trapezoidal rule by the sum of the areas between each chronological pair of assessments (using observed times). The weighted mean was then determined by dividing the AUC by the observed length of the collection interval (time of last assessment - time of first assessment in h). Analysis was done using analysis of covariance (ANCOVA) model where, change from baseline was summation of baseline, period, sequence and treatment. Participants were fitted as a random effect.
Time Frame: Baseline (Day -1) and Day 7 of each treatment period
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/deciliter
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 12 | 14
mg/deciliter
  Fasting Value | -12.325 (36.1277) | 7.479 (44.6181)
  Maximum (0-4 h) | 6.250 (45.2270) | 22.857 (49.1307)
  Maximum (4-10 h) | -6.583 (45.4402) | 29.714 (42.1251)
  Maximum (10-14 h) | 2.500 (51.34819) | 40.307 (56.18196)
  Maximum (0-24 h) | 4.583 (45.9020) | 23.071 (39.6959)
  AUC (0-4 h) Weighted Mean | 6.0737 (43.37336) | 22.0247 (46.54980)
  AUC (4-10 h) Weighted Mean | -4.6051 (43.31083) | 24.7262 (39.21502)
  AUC (10-14 h) Weighted Mean | 4.4221 (55.00201) | 38.2479 (51.91011)
  AUC (0-24 h) Weighted Mean | -2.0829 (44.76645) | 26.0704 (40.74711)
Statistical Analysis 1: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for Fasting Value; Test type: Superiority or Other; Mean Difference (Net) = -28.13, 95% CI 2-sided [-50.40 to -5.86] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for Fasting Value
Statistical Analysis 2: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for Maximum (0-4 h) Value; Test type: Superiority or Other; Mean Difference (Net) = -29.16, 95% CI 2-sided [-51.68 to -6.64] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for Maximum (0-4 h) Value
Statistical Analysis 3: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for Maximum (4-10 h) Value; Test type: Superiority or Other; Mean Difference (Net) = -36.58, 95% CI 2-sided [-62.25 to -10.90] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for Maximum (4-10 h) Value
Statistical Analysis 4: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for Maximum (10-14 h) Value; Test type: Superiority or Other; Mean Difference (Net) = -45.41, 95% CI 2-sided [-72.80 to -18.03] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for Maximum (10-14 h) Value
Statistical Analysis 5: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for Maximum (0-24 h) Value; Test type: Superiority or Other; Mean Difference (Net) = -29.35, 95% CI 2-sided [-50.84 to -7.86] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for Maximum (0-24 h) Value
Statistical Analysis 6: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for AUC (0-4 h) Weighted Mean; Test type: Superiority or Other; Mean Difference (Net) = -26.14, 95% CI 2-sided [-45.80 to -6.49] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for AUC (0-4 h) Weighted Mean
Statistical Analysis 7: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for AUC (4-10 h) Weighted Mean; Test type: Superiority or Other; Mean Difference (Net) = -32.00, 95% CI 2-sided [-55.41 to -8.58] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for AUC (4-10 h) Weighted Mean
Statistical Analysis 8: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for AUC (10-14 h) Weighted Mean; Test type: Superiority or Other; Mean Difference (Net) = -40.96, 95% CI 2-sided [-66.64 to -15.29] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for AUC (10-14 h) Weighted Mean
Statistical Analysis 9: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Treatment A-GSK2330672 + Metformin versus Treatment B-Placebo + Metformin for AUC (0-24 h) Weighted Mean; Test type: Superiority or Other; Mean Difference (Net) = -34.76, 95% CI 2-sided [-54.67 to -14.85] — The point estimate was calculated as least square mean difference (net values) of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for AUC (0-24 h) Weighted Mean

14. Secondary Outcome: AUC From Time 0 to 10 h (AUC 0-10 h) of Metformin in Presence of GSK2330672 or Placebo on Day 7
Description: AUC(0-10) for metformin when co-dosed with GSK2330672 or placebo is defined as the the area under the plasma concentration-time curve from time 0 to 10 h. It was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples were collected at 0 h (pre-dose within 15 min of dose and began eating breakfast immediately after taking study drug and finished eating in 15 min), 0.25 h, 0.50 h, 1 h, 2 h, 3 h, 4 h (pre-lunch), 5 h, 5.5 h, 6 h, 8 h and 10 h (pre-dinner) on Day 7. Analysis was done using a mixed effects model with fixed effect terms for treatment, period, and sequence. Participant within sequence was fitted as a random effect in the model.
Time Frame: Pre-dose (0 h), 0.25 h, 0.50 h, 1 h, 2 h, 3 h, 4 h (pre-lunch), 5 h, 5.5 h, 6 h, 8 h and 10 h (pre-dinner) on Day 7 of each treatment period
Population: Pharmacokinetic (PK) Population was defined as participants from the safety population who had plasma metformin and or GSK2330672 PK parameter estimates from any portion of the study. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram (ng)*h/mL
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 12 | 14
Nanogram (ng)*h/mL | 9189.2649 (34.080) | 9232.5372 (24.404)
Statistical Analysis 1: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Test type: Superiority or Other; Ratio = 1.013, 90% CI 2-sided [0.912 to 1.125] — The point estimate was calculated as geometric least square mean ratio of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for AUC (0-10 h)

15. Secondary Outcome: Maximum Plasma Concentration of Metformin (Cmax) in Presence of GSK2330672 or Placebo on Day 7
Description: Cmax is defined as the first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data Blood samples were collected at 0 h (pre-dose within 15 min of dose and began eating breakfast immediately after taking study drug and finished eating in 15 min), 0.25 h, 0.50 h, 1 h, 2 h, 3 h, 4 h (pre-lunch), 5 h, 5.5 h, 6 h, 8 h and 10 h (pre-dinner) on Day 7. Analysis was done using a mixed effects model with fixed effect terms for treatment, period, and sequence. Participant within sequence was fitted as a random effect in the model.
Time Frame: as for outcome 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 12 | 14
ng/mL | 1707.1 (28) | 1638.3 (25)
Statistical Analysis 1: Comparison: Treatment A-GSK2330672 + Metformin vs Treatment B-Placebo + Metformin; Test type: Superiority or Other; Ratio = 1.036, 90% CI 2-sided [0.937 to 1.145] — The point estimate was calculated as geometric least square mean ratio of Treatment A-GSK2330672 + Metformin and Treatment B-Placebo + Metformin for Cmax

16. Secondary Outcome: Median Time to Observed Peak Plasma Concentration (Tmax) When Co-dosed With GSK2330672 or Placebo on Day 7
Description: Tmax is defined as the time at which Cmax is observed, determined directly from the raw concentration-time data. Blood samples were collected at 0 h (pre-dose within 15 min of dose and began eating breakfast immediately after taking study drug and finished eating in 15 min), 0.25 h, 0.50 h, 1 h, 2 h, 3 h, 4 h (pre-lunch), 5 h, 5.5 h, 6 h, 8 h and 10 h (pre-dinner) on Day 7.
Time Frame: as for outcome 14
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
Number analyzed (Participants) | 12 | 14
h | 1.4583 [0.500 to 2.000] | 1.0000 [1.000 to 2.000]

ADVERSE EVENTS:
Time Frame: AE's and SAE's were collected from the start of study treatment of metformin in the run-in period and until Follow-up (up to 53 days)
Description: Safety Population was used.
Arm/Group | Treatment A-GSK2330672 + Metformin | Treatment B-Placebo + Metformin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 12/14 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A-GSK2330672 + Metformin (N=14) | Treatment B-Placebo + Metformin (N=14)
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A-GSK2330672 + Metformin (N=14) | Treatment B-Placebo + Metformin (N=14)
Diarrhoea (Gastrointestinal disorders) | 11 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.